CLINICAL TRIAL: NCT07130461
Title: Three-Dimensional Computed Tomography Assessment of Arcuate Foramen Variants and Their Surgical Implications: A Retrospective Observational Study
Brief Title: Prevalence and Surgical Implications of the Arcuate Foramen: A 3D CT-Based Observational Study
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilke Tamdogan, Assistant Professor, Ondokuz Mayıs University
Other Study IDs: E-53593568-771-250207806
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Arcuate Foramen; Anatomical Variations; Spine Surgery Complications
Keywords: Arcuate Foramen; 3D Computed Tomography; Vertebral Artery; Volume Rendering; OsiriX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Adults Undergoing Head CT/CTA (2023-2025): Consecutive adult patients (≥18 years) whose high-quality 3D CT or CTA images included the atlas (C1) vertebra. Images were evaluated retrospectively for the presence, type (complete/incomplete), and laterality (right/left/bilateral) of the arcuate foramen.

SUMMARY:
This study aims to determine the prevalence and types of the arcuate foramen (AF), an anatomical variation of the first cervical vertebra (atlas), using three-dimensional computed tomography (3D CT). The arcuate foramen is formed when a bony bridge develops over the groove for the vertebral artery. Although often asymptomatic, it may increase the risk of vascular or nerve injury during surgery in the craniovertebral junction region.

In this retrospective observational study, 3D CT scans of 200 adult patients obtained between January 2023 and July 2025 at Giresun University Faculty of Medicine were reviewed. The presence of AF was classified as complete or incomplete, and also categorized according to its location (right, left, or bilateral). Associations with demographic variables (age, sex) were analyzed.

The results will help improve awareness of AF in preoperative planning for neurosurgical and spinal procedures, potentially reducing the risk of complications involving the vertebral artery and surrounding neurovascular structures.

DETAILED DESCRIPTION:
The arcuate foramen (AF) is an anatomical variation of the atlas (C1 vertebra) that occurs when a bony bridge forms over the groove for the vertebral artery, creating a complete or partial tunnel. While frequently asymptomatic, its presence has been associated with conditions such as vertebrobasilar insufficiency, cervicogenic headache, and chronic neck pain. Importantly, AF may alter the course of the vertebral artery and suboccipital nerve, increasing the risk of injury during craniovertebral junction surgery, C1-C2 instrumentation, and posterior fossa approaches.

This retrospective cross-sectional study reviewed 3D computed tomography (CT) images of 200 adult patients obtained between January 2023 and July 2025 at Giresun University Faculty of Medicine. Images were reconstructed and analyzed using OsiriX MD software with a 3D volume rendering technique. AF was classified as complete or incomplete and further categorized by side (right, left, or bilateral). Associations with demographic variables, including age and sex, were examined.

Prevalence estimates were calculated with 95% confidence intervals. Interobserver agreement between two experienced neurosurgeons was assessed using Cohen's Kappa statistic. The findings aim to provide a clearer understanding of AF prevalence in the Turkish population and its potential surgical relevance. By identifying these variations preoperatively, surgeons can better plan instrumentation trajectories and minimize neurovascular complications in craniovertebral and upper cervical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of imaging
* High-quality CT or CTA images including the atlas (C1) vertebra and posterior arch
* Imaging obtained between January 2023 and July 2025 at Giresun University Faculty of Medicine
* Images suitable for 3D volume rendering analysis without significant artifacts

Exclusion Criteria:

* Motion or metallic artifact preventing adequate evaluation of atlas anatomy
* Prior cervical spine surgery or trauma affecting the atlas
* Congenital anomalies or severe deformity of the atlas obscuring posterior arch assessment
* Incomplete demographic or imaging data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) who underwent head computed tomography (CT) or computed tomography angiography (CTA) at Giresun University Faculty of Medicine between January 2023 and July 2025, whose images included the atlas (C1) vertebra and met quality criteria for three-dimensional reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of Arcuate Foramen Variants | Baseline (single review of existing imaging data)
  Proportion of participants with complete arcuate foramen identified on 3D computed tomography (CT).
  Unit of Measure: Percentage (%) of participants.
  Measurement Tool: High-resolution 3D reconstructed craniovertebral junction CT images, evaluated independently by two neuroradiologists.
  Analysis: Proportion calculated with 95% confidence intervals (CI).

SECONDARY OUTCOMES:
Association between Arcuate Foramen Type and Demographic Characteristics (Age and Sex) | Baseline.
  Description: Relationship between arcuate foramen type (complete vs. incomplete) and patient demographics, including age and sex distribution.
  Unit of Measure:
  Age: Mean ± standard deviation (years)
  Sex: Percentage (%) of male and female participants
  Measurement Tool: Demographic data (age and sex) recorded from electronic medical records.
  Analysis:
  Age: Independent t-test or Mann-Whitney U test; effect size with 95% confidence interval (CI).
  Sex: Chi-square test or Fisher's exact test; odds ratio (OR) with 95% CI.
  Unit of Measure: Mean ± standard deviation (years).
  Measurement Tool: Age recorded from electronic medical records.
  Analysis: Independent t-test or Mann-Whitney U test; effect size with 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Tamdogan, MD, Principal Investigator — Giresun University Faculty of Medicine
Locations (1):
- Giresun University Faculty of Medicine, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study involves retrospective analysis of de-identified radiological images. Individual participant data will not be shared to protect patient confidentiality.

REFERENCES:
- [Result] Arslan D, Ozer MA, Govsa F, Kitis O. The Ponticulus Posticus as Risk Factor for Screw Insertion into the First Cervical Lateral Mass. World Neurosurg. 2018 May;113:e579-e585. doi: 10.1016/j.wneu.2018.02.100. Epub 2018 Feb 25. PMID 29486308
- [Result] Pekala PA, Henry BM, Pekala JR, Hsieh WC, Vikse J, Sanna B, Walocha JA, Tubbs RS, Tomaszewski KA. Prevalence of foramen arcuale and its clinical significance: a meta-analysis of 55,985 subjects. J Neurosurg Spine. 2017 Sep;27(3):276-290. doi: 10.3171/2017.1.SPINE161092. Epub 2017 Jun 16. PMID 28621616
- [Result] Elliott RE, Tanweer O. The prevalence of the ponticulus posticus (arcuate foramen) and its importance in the Goel-Harms procedure: meta-analysis and review of the literature. World Neurosurg. 2014 Jul-Aug;82(1-2):e335-43. doi: 10.1016/j.wneu.2013.09.014. Epub 2013 Sep 18. PMID 24055572

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-31): https://cdn.clinicaltrials.gov/large-docs/61/NCT07130461/Prot_SAP_000.pdf